CLINICAL TRIAL: NCT07384156
Title: Enhancing Orthographic Communication and Literacy Outcomes for AAC Learners: Investigating Effective Instructional Strategies
Brief Title: Enhancing Orthographic Communication and Literacy Outcomes for AAC Learners
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jessica Caron, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 251267
Record Dates: First submitted 2026-01-23; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Literacy; Communication, Nonverbal
Keywords: literacy; augmentative and alternative communication; nonverbal; Communication; Autism; Intellectual Disabilities
MeSH Terms: conditions — Literacy; Nonverbal Communication; Communication; Autistic Disorder; Intellectual Disability

STUDY DESIGN:
Intervention Model Description: 30 children will receive ALLSTAR - SC (standard use of ALLSTAR) and 30 children will receive ALLSTAR - I (integrated approach)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALLSTAR-SC (Active Comparator): The ALL app comes with lessons in early literacy skills, with the materials are pre-made, and tasks are modified to support independent participation by AAC users. By using ALLSTAR as "Standard of Care", the evidence base has the potential to increase by demonstrating related to demonstration that AAC users can learn multiple skills and when provided the opportunity to learn phonics. Intervention with the app includes 50 trials per lesson and an instructional sequence that service providers are trained to implement, including: introducing the skill, two model trials, five trials using guided practice techniques, and three trials of independent practice with corrective feedback. The words and skills will rotate based on lesson number and the automated data collected within the technology. The AAC user will get exposure to four skills per lesson.
  Interventions: Behavioral: ALLSTAR
- ALLSTAR-I* (Experimental): In ALLSTAR-I* condition, this group will receive explicit instruction in encoding and phoneme-grapheme knowledge, adding an integrative decoding and encoding approach within the lessons. Studies have shown that combining instruction on phonological awareness and letter-sound correspondences with word reading and spelling better develops students' word reading and spelling skills. These integrated lessons will be incorporated starting at lesson 20 and will include the features based on a refined intervention including the "Hear, Say, Type, Read, Use" strategy.
  Interventions: Behavioral: ALLSTAR

INTERVENTIONS:
Behavioral: ALLSTAR — The ALL app comes with lessons in early literacy skills, with three tiers of lessons available. Both intervention groups will use ALLSTAR materials, including an implementation binder and the ALL app. Both intervention groups will also receive daily instruction by a trained service provider (~30 mins. Per day). Additionally, in support of best practices, both groups will receive phonics instruction and use of explicit and systematic instruction for four skills per day and 50 trials per lesson. Lessons will differ based on skills targeted.

SUMMARY:
The goal of this clinical trial is to determine whether adding Integrated Decoding and Encoding instruction to the ALLSTAR literacy program improves reading outcomes for students with significant literacy and communication needs. The study will also examine how students' reading skills change over time across instructional conditions.

The main questions it aims to answer are:

Do students who receive ALLSTAR with Integrated Decoding and Encoding instruction demonstrate greater improvements in literacy outcomes than students who receive ALLSTAR as standard care alone? How do students' literacy skills change from baseline to mid-intervention and post-intervention across the two instructional conditions? Researchers will compare two groups using a randomized controlled trial design. One group will receive 60 lessons of ALLSTAR as the standard of care (ALLSTAR-SC), and the other group will receive 60 lessons of ALLSTAR with the addition of Integrated Decoding and Encoding lessons (ALLSTAR-I*). Literacy outcomes will be measured using repeated assessment probes at baseline (0 Lessons), after 30-40 lessons, and after 60 lessons to evaluate differences between groups and changes over time in the individuals.

DETAILED DESCRIPTION:
Literacy skills enhance public health outcomes (employment, safety, well-being, and social engagement). Additionally and critically, for individuals who cannot speak and use augmentative and alternative communication (AAC; pointing to pictures, using a speech generating device), literacy skills support precise communication by allowing individuals to spell the exact words they wish to communicate. However, over 90% of AAC users leave high school illiterate. The long-term goal for this project is improve language and literacy outcomes in individuals who use AAC, consequently improving health and well-being outcomes. While recent research underscores the importance of explicit literacy instruction that integrates decoding and encoding, encoding is rarely taught to AAC users, and it is not yet known if this approach will yield better language and literacy outcomes among AAC users. The focus of the current proposal is to teach decoding and encoding using an integrated approach to instruction with an existing literacy curriculum, ALLSTAR. ALLSTAR and approaches using the ALL app have resulted in learning across all AAC users, with large to very large effect sizes observed (Tau-U ranges: .63 - 1.0) and large gains (+44% on pre-post ELA assessment).

The project goal is to: (1) adapt and evaluate the effect of an integrated approach in an AAC literacy intervention on CVC decoding and encoding using an iterative single subject design; (2) evaluate the effect of adding the integrated "spell-to-read" approach to ALLSTAR using an RCT (N=60); and (3) assess the acceptability, feasibility, and adoptability of the literacy lessons by practitioners, in order to understand the barriers and facilitators that influence their uptake, ultimately increasing the use of evidence-based literacy instruction for AAC users. Data measurements related to the respective aims above, include: (1) percent gains and intervention effectiveness, (2) gains on Pre, Mid, and Post scores on Early Literacy Assessment (letter-sounds, sound blending, phoneme segmentation, decoding, irregular sight words, and encoding); and (3) thematic analysis and scores on the Feasibility Adoption Acceptability Questionnaire (FAAQ), completed at three timepoints throughout each study. Our expected outcome is the development of an effective and adoptable literacy intervention for children who use AAC.

The significance of this work is that it will advance a new intervention paradigm for AAC users that capitalizes on an explicit connection between literacy and communication to foster AAC users who can communicate orthographically and ultimately more precisely what they wish to express. This proposal is timely, in that it is responsive to NIDCD's mission and responsive to and collaborative with AAC users. The project has the potential for high clinical impact in changing poor literacy outcomes for a population that is unjustly denied evidence-based literacy instruction.

ELIGIBILITY:
Inclusion Criteria:

* Have complex communication needs and use AAC,
* are ages 5-12,
* per report can follow two-step directions,
* symbolic communicators with at least 75 words on the CDI and mean length of utterance greater than 2
* can match letters and words with greater than 90% accuracy,
* can identify letter-sound correspondences from a field of 4 with greater than 70% accuracy
* can identify common photographs used to represent words in the study (e.g., touch the picture of a hat, touch hot) with greater than 80% accuracy,
* can sit to work in a minimum of 5 min. intervals
* decoding or encoding at less than 40% accuracy based on parent or provider report and screening results;
* demonstrate functional vision and hearing

Exclusion Criteria:

* • Do not have complex communication needs / can speak and do not need AAC,

  * Younger than 5 or older than 12 years of age,
  * Can not follow two-step directions,
  * Are not symbolic communicators with at least 75 words on the CDI and not combining at least 2 symbols
  * Can not match letters and words with >90% accuracy,
  * Can not identify letter-sound correspondences from a field of 4 with greater than 70% accuracy
  * Can not identify common photographs used to represent words in the study (e.g., touch the picture of a hat, touch hot) with greater than 80% accuracy,
  * Can not attend to work for 5 mins.
  * decoding or encoding at more than 40% accuracy based on parent or provider report and screening results;
  * Do not have corrected or functional vision and hearing

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Percent correct on Early Literacy Assessment (ELA) | At study completion of the required 60 lessons, an average of 5 months
  Early Literacy Assessment (ELA) is a 120 question measure that covers six literacy skills. It was specifically created for a population with minimal or no speech. The ELA will be used to assess progress in domains of: letter-sound correspondence, sound blending, decoding, grapheme-phoneme typing, and encoding.

SECONDARY OUTCOMES:
The difference between the two literacy interventions for individuals who have minimal or no speech | After study completion, an average of 5 months
  Scores from the Early Literacy Assessment (ELA) will be analyzed in this secondary outcome measure to look at the difference between the two interventions. The ELA has 120 questions. The total scores on ELA between the two interventions will be compared using independent t-tests and Cohens D.

OTHER OUTCOMES:
Qualitative Analysis of Service Provider's Social Validity of the two literacy interventions | Three times through the course of the study, on average at 0, 10, and 20 weeks.
  To measure the perceptions of implementation variables, a Feasibility Adoption Acceptability Questionnaire (FAAQ) will be completed. The FAAQ was used in our pilot studies and was developed based on the Evidence-Based Practice Attitude Scale (EBPAS). The FAAQ includes 8 Likert questions and 2 open-ended questions. The Qualitative analysis of these will help supporting understanding of acceptability, adoption, sustainment, and feasibility of the two literacy interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared. IPD will include de-identified survey and questionnaire responses, coded interview data (themes only, with no direct identifiers), and analyzable outcome data such as pre-post measures of decoding, encoding, and English Language Arts (ELA) performance (e.g., scores and percentage gains). No information that could reasonably identify individual participants will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: De-identified IPD will be made publicly available through the Open Science Framework (OSF; https://osf.io) in open-access formats (e.g., Excel or CSV files). Data will be accessible without restriction to researchers and the public. The data will be available beginning after publication of the primary study results and will remain available indefinitely. A direct link to the OSF repository will be provided in the ClinicalTrials.gov record in the Available IPD/Information field once the data are posted.
URL: https://osf.io